CLINICAL TRIAL: NCT06356532
Title: the Effectiveness of the Intensive Care Unit Diary for Intensive Care Unit Liver Transplant Recipients
Brief Title: the Intensive Care Unit Diary for Liver Transplant Recipients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202312197544
Record Dates: First submitted 2024-03-30; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-03

CONDITIONS: Liver Transplant Disorder

STUDY DESIGN:
Intervention Model Description: The participants in the control group received the routine care including communication and companionship provided by the nurses of the intensive care unit.
  The participants in the intervention group received the intensive care unit diary writing and reading. Participants are required to write at least one sentence daily. The primary writers will be the patients themselves, and in cases where patients are unable to write, their family members will write on their behalf. After completion, the diary will be handed over to the patients to review its contents for at least 10 minutes before bedtime, allowing them to write down their immediate reflections and thoughts on when they read. This process will continue until the 14th day post-operation.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor is blinded to the group assignments of the patients. She is tasked with collecting the measured outcomes from the patients. Data collection will be conducted by co-principal investigator of the research team. She will distribute the questionnaires at enrollment, and on the 7th and 14th days post-operation. Once notified by the researchers, data collector will distribute and collect the questionnaires. Upon completion, the questionnaires will be sealed in envelopes by the data collectors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The participants in the intervention group received the intensive care unit diary writing and reading. Participants are required to write at least one sentence daily. The primary writers will be the patients themselves, and in cases where patients are unable to write, their family members will write on their behalf. After completion, the diary will be handed over to the patients to review its contents for at least 10 minutes before bedtime, allowing them to write down their immediate reflections and thoughts on when they read. This process will continue until the 14th day post-operation.
  Interventions: Behavioral: intensive care unit diary
- control group (No Intervention): The participants in the control group received the routine care including communication and companionship provided by the nurses of the intensive care unit.

INTERVENTIONS:
Behavioral: intensive care unit diary — The intensive care unit diary is a notebook provided to patients during their stay in the intensive care unit, allowing them to record all events that occur during this period. Patients are encouraged to freely write about their experiences, which may include details about their treatment progress, daily activities, visits from family members, and other relevant aspects of their stay.
  Arms: experimental group

SUMMARY:
the purpose of this study is to assess the effectiveness of the intensive care unit diary for intensive care unit liver transplant recipients.

DETAILED DESCRIPTION:
This study was a prospective two-armed randomized clinical trial to assess the effectiveness of the intensive care unit diary for intensive care unit liver transplant recipients. The investigators used simple random allocation with a drawing from a lots container to divide the sample into an experimental group and a control group. The participants in the control group received the routine care including communication and companionship provided by the nurses of the intensive care unit. The participants in the intervention group received the intensive care unit diary writing and reading. Participants are required to write at least one sentence daily. The primary writers will be the patients themselves, and in cases where patients are unable to write, their family members will write on their behalf. After completion, the diary will be handed over to the patients to review its contents for at least 10 minutes before bedtime, allowing them to write down their immediate reflections and thoughts on when they read. This process will continue until the 14th day post-operation.

There will be a total of three time questionnaire, each taking 10-15 minutes to complete. The first questionnaire will be administered upon enrollment and will include self-constructed basic demographic and disease-related attribute questionnaires, Depression-Anxiety-Stress scale, Brief Symptom Rating Scale , and a Sense of Coherence Scale. The second questionnaire will be administered on the 7th day post-operation, consisting of Depression-Anxiety-Stress scale, Brief Symptom Rating Scale , and a Sense of Coherence Scale. The third questionnaire will be administered on the 14th day post-operation, containing Depression-Anxiety-Stress scale, Brief Symptom Rating Scale , and a Sense of Coherence Scale.Data collection will be conducted by co-principal investigator of the research team. She will distribute the questionnaires at enrollment, and on the 7th and 14th days post-operation. Once notified by the researchers, data collector will distribute and collect the questionnaires. Upon completion, the questionnaires will be sealed in envelopes by the data collectors. The data will be analyzed to investigate the effectiveness of the intervention in reducing stress, depression, and anxiety in liver transplant patients, as well as sense of coherence and reducing the incidence of delirium.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to sign the written informed consent form.
* Admission to the intensive care unit for liver transplant surgery.
* Ability to read and write in Chinese and communicate in either Chinese or Taiwanese dialect.
* Adults aged 18 years or older, both male and female.

Exclusion Criteria:

* Diagnosis of a mental illness.
* Presence of intellectual, cognitive, or hearing impairments.
* Use of sedative medications and scoring less than -2 on the Richmond Agitation-Sedation Scale (RASS).
* Inability of family members to visit during the patient's stay in the intensive care unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
change from baseline in depression on the Depression-Anxiety-Stress scale at post operation day 7 and day 14 | Baseline and post operation day 7 and day 14
  The Depression-Anxiety-Stress scale is a validated, self reported instrument assessing depression over the past 7days period. Possible scores range from 0 (no depression)-21 (worst depression).
  Change=( post operation day 7 score-Baseline score)&( post operation day 14 score-Baseline score)
change from baseline in anxiety on the Depression-Anxiety-Stress scale at post operation day 7 and day 14 | Baseline and post operation day 7 and day 14
  The Depression-Anxiety-Stress scale is a validated, self reported instrument assessing anxiety over the past 7days period. Possible scores range from 0 (no anxiety)-21 (worst anxiety).
  Change=( post operation day 7 score-Baseline score)&( post operation day 14 score-Baseline score)
change from baseline in stress on the Depression-Anxiety-Stress scale at post operation day 7 and day 14 | Baseline and post operation day 7 and day 14
  The Depression-Anxiety-Stress scale is a validated, self reported instrument assessing stress over the past 7days period. Possible scores range from 0 (no stress)-21 (worst stress).
  Change=( post operation day 7 score-Baseline score)&( post operation day 14 score-Baseline score)
change from baseline in sense of coherence on the Sense of Coherence Scale at post operation day 7 and day 14 | Baseline and post operation day 7 and day 14
  The Sense of Coherence Scale is a validated, self reported instrument assessing sense of coherence. Possible scores range from 0 (worst)-91(best).
  Change=( post operation day 7 score-Baseline score)&( post operation day 14 score-Baseline score)
change from baseline in emotional stress on the Brief Symptom Rating Scale at post operation day 7 and day 14 | Baseline and post operation day 7 and day 14
  The Brief Symptom Rating Scale is a validated, self reported instrument assessing emotional distress. Possible scores range from 0 (best)-15(worst).
  Change=( post operation day 7 score-Baseline score)&( post operation day 14 score-Baseline score)

SECONDARY OUTCOMES:
change from baseline in delirium on the intensive care delirium screening checklist at post operation day 1 and day 14 | post operation day 1 and day 14
  The the intensive care delirium screening checklist is a validated instrument assessing delirium. Possible scores range from 0 (best)-8(worst).
  Change=( post operation day 14 score-post operation day 1 score)

CONTACTS AND LOCATIONS:
Overall Officials: Jyun-Sian WU, Master, Study Chair — Chang Gung Memorail Hospital

IPD SHARING:
Plan to Share IPD: No